CLINICAL TRIAL: NCT03976700
Title: Bufei Jianpi Granule for Delaying Pulmonary Function Decline in Early-Stage COPD: A Randomized, Double-blind, Placebo Controlled Trial
Brief Title: Bufei Jianpi Granule for Delaying Pulmonary Function Decline in Early-Stage COPD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Collaborators: Jiangsu Province Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCM for Early-Stage COPD
Record Dates: First submitted 2019-05-29; First posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Bufei Jianpi Granule; Randomized Controlled Trial
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bufei Jianpi granule (Experimental): Patients in this arm will receive Bufei Jianpi granule.
  Interventions: Drug: Bufei Jianpi granule
- Placebo Bufei Jianpi granule (Placebo Comparator): Patients in this arm will receive placebo Bufei Jianpi granule.
  Interventions: Drug: Placebo Bufei Jianpi granule

INTERVENTIONS:
Drug: Bufei Jianpi granule — Bufei Jianpi granule is composed of many kinds of traditional Chinese medicine. The granule will be administered twice daily for five days a week for 104 weeks.
  Arms: Bufei Jianpi granule
Drug: Placebo Bufei Jianpi granule — Placebo Bufei Jianpi granule consists of dextrin, bitter and 5% of the Bufei Jianpi granule. The appearance, weight, color and odor of the preparation are the same as those of treatment group. The placebo granule will be administered twice daily for five days a week for 104 weeks.
  Arms: Placebo Bufei Jianpi granule

SUMMARY:
This study aims to establish the treatment scheme of Bufei Jianpi granule for early-stage (GOLD stage 1 or 2) chronic obstructive pulmonary disease (COPD), delaying pulmonary function decline and forming high quality evidence.

DETAILED DESCRIPTION:
COPD is a highly prevalent disease, with a prevalence among people 40 years of age or older of 10.1% worldwide and 13.7% in China. COPD has become the third leading cause of death worldwide. More than 70% of patients with COPD are in GOLD stage 1 (mild) or 2 (moderate), with very mild or no apparent respiratory symptoms such as dyspnea. The Tiotropium in Early Chronic Obstructive Pulmonary Disease Patients in China (Tie-COPD) trial was designed to investigate the effect of tiotropium on the FEV1 in COPD patients with GOLD stage 1 or 2. The investigator's previous studies also suggested that traditional Chinese medicine (TCM) has effect on GOLD stage 1 or 2 COPD.

This is a multicenter, randomized, double-blind, placebo controlled trial to evaluate the effect of Bufei Jianpi granule for delaying pulmonary function decline in early-stage (GOLD stage 1 or 2) COPD subjects. After a 14-day run-in period, 612 subjects will be randomly assigned to treatment group or control group for 104-week treatment. The primary outcomes include pulmonary function and frequency of acute exacerbation. The secondary outcomes include clinical symptoms, dyspnea, exercise capacity, quality of life and treatment satisfaction. Safety will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of early-stage (GOLD stage 1 or 2) COPD.
* Syndrome differentiation meets criteria of Qi deficiency of the lung syndrome, Qi deficiency of the lung and spleen syndrome or Qi deficiency of the lung and kidney syndrome.
* Age ranges from 40 years to 80 years.
* With informed consent signed.

Exclusion Criteria:

* Pregnant and lactating women.
* Patients with severe cardiovascular and cerebrovascular diseases.
* Patients with severe liver and kidney diseases.
* Patients with asthma, bronchiectasis, active pulmonary tuberculosis, pulmonary embolism or other severe respiratory diseases.
* Patients with tumor after resection, radiotherapy or chemotherapy in the past 5 years.
* Patients with severe neuromuscular disorders, severe arthritis or severe peripheral vascular diseases.
* Patients with severe cognitive and psychiatric disorders.
* Patients with diabetes.
* People who are allergic to the treatment drugs.
* Patients who have participated in other clinical studies in the past 4 weeks.
* Patients who have experienced one or more acute exacerbation in the past 4 weeks.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
FEV1 | Change from baseline FEV1 at week 26, 52, 78 and 104.
  Forced expiratory volume in one second ( FEV1) will be used to assess pulmonary function.
Frequency of acute exacerbation | Up to week 104.
  Frequency of acute exacerbation will be recorded.

SECONDARY OUTCOMES:
Clinical symptom assessment questionnaire | Change from baseline clinical symptom assessment questionnaire scores at week 13, 26, 39, 52, 65, 78, 91 and 104.
  Clinical symptom assessment questionnaire of COPD will be used to assess symptom.
mMRC | Change from baseline mMRC scores at week 13, 26, 39, 52, 65, 78, 91 and 104.
  The modified Medical Research Council dyspnoea scale (mMRC) will be used to assess severity of dyspnea.
6MWD | Change from baseline 6MWD at week 13, 26, 39, 52, 65, 78, 91 and 104.
  Six-minute walk distance (6MWD) will be conducted to assess exercise capacity.
CAT | Change from baseline CAT scores at week 13, 26, 39, 52, 65, 78, 91 and 104.
  The COPD assessment test (CAT) is a self-administered questionnaire that measures health-related quality of life.
SF-36 | Change from baseline SF-36 scores at week 13, 26, 39, 52, 65, 78, 91 and 104.
  The MOS 36-Item Short-Form Health Survey (SF-36) will be used to assess quality of life.
mCOPD-PRO | Change from baseline mCOPD-PRO scores at week 13, 26, 39, 52, 65, 78, 91 and 104.
  The modified COPD patient-reported outcome scale (mCOPD-PRO) will be used to assess quality of life. The mCOPD-PRO contains 27 items in three domains. mCOPD-PRO scores range from 0 to 4 with a decrease in score showing higher health status.
EQ-5D | Change from baseline EQ-5D scores at week 13, 26, 39, 52, 65, 78, 91 and 104.
  EuroQol 5D (EQ-5D) will be used to assess quality of life.
mESQ-COPD | Change from baseline mESQ-COPD scores at week 13, 26, 39, 52, 65, 78, 91 and 104.
  The modified effectiveness satisfaction questionnaire for COPD (mESQ-COPD) will be used to assess treatment satisfaction. The mESQ-COPD contains 19 items in four domains. mESQ-COPD scores range from 0 to 4 with a decrease in score showing higher treatment satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Jiansheng Li, Professor, Study Chair — The First Affiliated Hospital of Henan University of Traditional Chinese Medicine
Locations (1):
- The First Affiliated Hospital of Henan University of Traditional Chinese Medicine, Zhengzhou, Henan, China